CLINICAL TRIAL: NCT04779632
Title: Fish Oil Affects Cognition and ADHD Symptoms in Adults With Autism Spectrum Disorder: A Randomized Crossover Study
Brief Title: Fish Oil Affects Cognition and ADHD Symptoms in Adults With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Professor Lotte Lauritzen, Professor Lotte Lauritzen, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D227
Record Dates: First submitted 2021-02-03; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Randomized 2 x 4 weeks head-to-tail crossover trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A person, who was not involved in the data collection generated the randomization list (online tool) and packed both types of capsules in containers of similar appearance and labeled them with ID and period. The participants were allotted to ID numbers based on date and time of their first visit and supplied with the relevant capsule container in the beginning of each period.
  The oil capsules were provided by two different companies and not the same size: 1 ml Eskimo-3 High 65% (Midsona Malmӧ, Sweden) and 0.75 ml SO (Natur-Drogeriet A/S, Hørning, Denmark). Containers were only handled by colleagues and participants and the investigator tried to prevent un-blinding due to differences in rattling sound by use of noise-cancelling in-ear headphones.
  Blinding was checked by asking the participants and the investigator to guess which oil they had received at the end of the interventions. Formal un-blinding did not occur before the primary statistical analyses was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crossover study: Fish Oil --> Safflower Oil (Other): 4 weeks of fish oil supplementation followed by 4 weeks of safflower oil supplementation
  Interventions: Dietary Supplement: Experimental: Fish Oil; Dietary Supplement: Comparator: Safflower Oil
- Crossover study: Safflower Oil --> Fish Oil (Other): 4 weeks of safflower oil supplementation followed by 4 weeks of fish oil supplementation
  Interventions: Dietary Supplement: Experimental: Fish Oil; Dietary Supplement: Comparator: Safflower Oil

INTERVENTIONS:
Dietary Supplement: Experimental: Fish Oil — Participants are provided with fish oil capsules and asked to take 4 capsules of 1000 mg twice a day (in total 5.2 mg/day of long-chain n-3 fatty acids hereof 2400 mg of eicosapentaenoic acid and 1600 mg of docosahexaenoic acid) for 4 weeks.
Dietary Supplement: Comparator: Safflower Oil — Participants are provided with fish oil capsules and asked to take 4 capsules of 500 mg twice a day (containing ~ 3000 mg of linoleic acid) for 4 weeks.

SUMMARY:
The prevalence of autism spectrum disorder (ASD) is rising and was estimated to have a prevalence of around 1.5% in developed countries in 2016. ASD is characterized by impairments in social interaction and repetitive behavior and is associated with executive dysfunction such as impaired working memory, inhibition, and flexibility. Furthermore, ASD is often associated with multiple comorbidities such as attention-deficit/hyperactivity disorder (ADHD), depression, and anxiety.

Systematic reviews and meta-analyses indicate that fish oil (FO) supplementation improves attention, impulsivity, and hyperactivity in children with ADHD and beneficial effects in adults with depression and anxiety. Some randomized trials in children with ASD have shown improvements on selected executive functions, but results from meta-analysis are inconsistent and no trial has examined the effect in adults with ASD. Furthermore, most of the previous studies have mainly assessed effects by questionnaires and no objective tests, only provided low doses (<1.5 g/d of n-3 long-chain polyunsaturated fatty acids) and none of them have examined the potential influence of comorbid ADHD, depression, or anxiety.

The aim of the study was to examine the effect of FO on sustained attention and visuospatial short-term memory memory, as well as cognitive inhibition, executive function, and core symptoms of ASD, and of ADHD, and social function in adults with ASD. In light of the shared and additive cognitive impairments in individuals with both ASD and ADHD, the hypothesis was that individuals with comorbid ADHD will show the most pronounced effects. The study furthermore aimed to examine potential interaction with depression, anxiety, and gender.

This was investigated in a randomized double-blind head-to-tail crossover trial in 26 adults with ASD, who are provided with FO and safflower oil (SO) for 4 weeks each. The subjects were examined at baseline and after each period with tests of attention and working memory (primary endpoints) as well as a test of cognitive flexibility and clinical questionnaires.

DETAILED DESCRIPTION:
The aim of the study was to examine the effect of fish oil (FO) on sustained attention and visuospatial short-term memory memory, as well as cognitive inhibition, executive function, and core symptoms of ASD, and of ADHD, and social function in adults with ASD. In light of the shared and additive cognitive impairments in individuals with both ASD and ADHD, the hypothesis was that individuals with comorbid ADHD will show the most pronounced effects. The study furthermore aimed to examine potential interaction with depression, anxiety, and gender.

This was investigated in a 2 × 4 week randomized double-blind head-to-tail crossover study with FO and safflower oil (SO).

Participants were recruited by advertisements posted in autism-related institutions and autism forums on Facebook as well as via personal networking. The study aimed to recruit up to thirty participants and ended up with twenty six participants.

The intervention in the two periods consisted of four capsules two times per day of FO (corresponding to approximately 5,2 g/d long-chain polyunsaturated fatty acids) and SO (1.2 g/day of linoleic acid), respectively. The intervention sequences: FO → SO or SO → FO was determined by a randomization list generated by a person, who was not involved in the data collection and FO and SO capsules were packed in white containers of similar appearance in the same known excess amount of what was required for four weeks. The participants were allotted to one of the intervention sequences by ID numbers based on date and time of their first visit and were provided with the appropriate pre-ID labelled container in the beginning of each period.

The participants were examined at baseline and after each period. The assessment consisted of the following: attention (The d2 Test of Attention) and spatial working memory (Corsi Block-Tapping Test) as primary outcomes and as secondary outcomes, inhibition and flexibility (The Stroop Word-Color Test), ADHD symptoms (Conners Rating Scale), and executive and social functions assessed by the Behavioral Inventory of Executive Function and Social Responsiveness Scale, respectively. Compliance was verified by whole-blood fatty acid analysis.

ELIGIBILITY:
Inclusion Criteria:

A clinical diagnosis of ASD (Asperger's syndrome, Autistic disorder, or a not otherwise specified pervasive developmental disorder).

Exclusion Criteria:

* Supplementation with n-3 long-chain polyunsaturated fatty acids 1 mo prior to the intervention or during the intervention.
* Major changes to psychopharmacological treatment 1 mo prior to the intervention or during the intervention.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Change in short-term spatial working memory | Baseline, 4 and 8 weeks
  Total Score (based on the total number of blocks in correct runs) in Corsi Block-Tapping Test (a higher is better)
Change in attention | Baseline, 4 and 8 weeks
  Total errors percent in d2-Test of Attention (d2-ToA): a measure of sustained attention

SECONDARY OUTCOMES:
Cognitive flexibility and inhibition | baseline, 4 and 8 weeks
  Reading time for color-word card (sec and relative to word and color card) in Stroop Color & Word Test (SCWT)
ADHD symptoms | baseline, 4 and 8 weeks
  The total symptoms score in Conners' Adult ADHD Rating Scale - Short: Self Report (CAARS - S:S) (range 0-54) including the subscores for attention (range 0-26) and hyperactivity/impulsivity (range 0-26) (higher scores are worse)
Executive function | baseline, 4 and 8 weeks
  The composite score in Behavioral Rating Inventory of Executive Function - Adult (BRIEF-A) (range 75-225) including the subscore for the metacognition index (range 45-135) and behavioral regulatory index (range 30-90) with focus on working memory, inhibition and flexibility from the two subscales, respectively (higher scores are worse)
ASD symptoms | baseline, 4 and 8 weeks
  The total score in Social Responsiveness Scale, Second Edition - Adult, Self-Report (SRS-2-ASR) (range 0-195) including the sub-scores for social communication and interaction (range for all sub-scores combined 0-159) and the score for repetitive behaviours and restricted interests (range 0-36) (higher scores are worse)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen - Department of Nutrition & Exercise, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No